CLINICAL TRIAL: NCT01137123
Title: A Prospective Clinical Trial of Improving the Treatment of Thoracic Esophageal Cancer
Brief Title: Improve the Treatment of Thoracic Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Peng Lin, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2007044
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2021-09

CONDITIONS: Thoracic Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- standard two field +follow-up (Active Comparator)
  Interventions: Procedure: standard two field Lymphadenectomy
- standard two field +adjuvant chemotherapy (Experimental)
  Interventions: Drug: adjuvant chemotherapy; Procedure: standard two field Lymphadenectomy
- total two field+follow-up (Experimental)
  Interventions: Procedure: Total two field Lymphadenectomy
- total two field+adjuvant chemotherapy (Experimental)
  Interventions: Drug: adjuvant chemotherapy; Procedure: Total two field Lymphadenectomy
- three field+follow-up (Experimental)
  Interventions: Procedure: three field Lymphadenectomy
- three field+adjuvant chemotherapy (Experimental)
  Interventions: Drug: adjuvant chemotherapy; Procedure: three field Lymphadenectomy

INTERVENTIONS:
Drug: adjuvant chemotherapy — Docetaxel 75mg/m2 +Nedaplatin 75mg/m2,IV drip on day 1 of each 21 day cycle. Number of cycles: till unacceptable toxicity develops and no more than 4 cycles.
  Arms: standard two field +adjuvant chemotherapy; three field+adjuvant chemotherapy; total two field+adjuvant chemotherapy
Procedure: standard two field Lymphadenectomy — Standard two field lymphadenectomy is standard mediastinal lymphadenectomy which defined by the International Association of esophageal disease(ISDE) of thoracic esophageal cancer.
  Other Names: two field(S)
  Arms: standard two field +adjuvant chemotherapy; standard two field +follow-up
Procedure: Total two field Lymphadenectomy — Total two field Lymphadenectomy is total mediastinal lymphadenectomy which defined by the International Association of esophageal disease(ISDE) of thoracic esophageal cancer.
  Other Names: two field(T)
  Arms: total two field+adjuvant chemotherapy; total two field+follow-up
Procedure: three field Lymphadenectomy — Three field Lymphadenectomy includes abdominal,mediastinal and cervical lymphadenectomy.
  Other Names: three field
  Arms: three field+adjuvant chemotherapy; three field+follow-up

SUMMARY:
The purpose of this study is

1. To compare the effects of the two types of thoracic esophageal cancer lymphadenectomy on the staging and prognosis of resectable esophageal cancer, which defined by the International Association of esophageal disease(ISDE) - standard mediastinal lymphadenectomy,total mediastinal lymphadenectomy and three field lymphadenectomy,and to find out reasonable range of lymphadenectomy.
2. To compare the effects of Chemotherapy Group (Docetaxel + Nedaplatin) with Control Group on the prognosis of resectable thoracic esophageal cancer,and to explore the indications of adjuvant chemotherapy.

DETAILED DESCRIPTION:
According to different location of the primary lesion，the subject can be allocated to two sub-groups:

The patient with upper or middle thoracic esophageal cancer may be assigned to two field(T)-total mediastinal lymphadenectomy group,which is control group in this study or three field lymphadenectomy-Abdominal + mediastinal + cervical lymphadenectomy group,which is study group in this study randomly.

After the operation,the patient whose primary lesion is completely(R0) resected will be assigned to adjuvant chemotherapy group or interview group randomly.

ELIGIBILITY:
Inclusion Criteria:

1. Age≤70 years old;
2. Karnofsky Performance Status（KPS）≥80;
3. Pathological diagnosis is squamous cell carcinoma of thoracic esophageal which is treated initially;
4. Clinical stage is c T 1 ~ 3 N 0 ~ 1 according to the results of endoscopic ultrasonography，chest and abdomen CT and neck ultrasonic.
5. The preoperative evaluation of organ function is tolerant of surgery and chemotherapy;
6. The subject can understand and sign the informed consent form (ICF);
7. The following laboratory tests, made in 4 weeks before first medication, confirmed that bone marrow, liver and kidney function in line with the requirements to participate in research; Hemoglobin（HGB）≥9.0g/L; absolute neutrophils count（ANC）≥1.5×109/L; platelet count（PLT）≥100×109/L; total bilirubin（TBIL）≤1.5N;aspartate aminotransferase (AST)≤2.5N;alanine aminotransferase(ALT)≤2.5N;prothrombin time(PT)≤1.5N, and activated partial thromboplastin time(APTT) is in normal range;endogenous creatinine clearance rate(CRE)≤1.5N.

Exclusion Criteria:

1. Cervical esophageal cancer and Non-squamous cell carcinoma of thoracic esophageal cancer;
2. Advanced Esophageal Cancer;
3. Prior malignancy in 5 years recently;
4. History of previous chest radiotherapy;
5. History of cardio-cerebral vascular accident in 6 months lately;
6. The subject can not understand and sign the informed consent form(ICF).

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2010-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
survival rate | 5 years
  1. Disease-free survival
  2. overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Peng Lin, Professor, Principal Investigator — 651, Dongfeng Road East, Guangzhou, P. R. China
Locations (1):
- Sun Yat-sen Uniersity Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Parkin DM, Bray FI, Devesa SS. Cancer burden in the year 2000. The global picture. Eur J Cancer. 2001 Oct;37 Suppl 8:S4-66. doi: 10.1016/s0959-8049(01)00267-2. No abstract available. PMID 11602373
- [Background] Urschel JD, Vasan H, Blewett CJ. A meta-analysis of randomized controlled trials that compared neoadjuvant chemotherapy and surgery to surgery alone for resectable esophageal cancer. Am J Surg. 2002 Mar;183(3):274-9. doi: 10.1016/s0002-9610(02)00795-x. PMID 11943125
- [Background] Peracchia A, Bonavina L, Ruol A, Stein H. Esophageal cancer: a European perspective. Recent Results Cancer Res. 2000;155:119-22. doi: 10.1007/978-3-642-59600-1_12. PMID 10693245
- [Background] Isono K, Sato H, Nakayama K. Results of a nationwide study on the three-field lymph node dissection of esophageal cancer. Oncology. 1991;48(5):411-20. doi: 10.1159/000226971. PMID 1745490
- [Background] Kato H, Watanabe H, Tachimori Y, Iizuka T. Evaluation of neck lymph node dissection for thoracic esophageal carcinoma. Ann Thorac Surg. 1991 Jun;51(6):931-5. doi: 10.1016/0003-4975(91)91008-j. PMID 2039322
- [Background] Nishihira T, Hirayama K, Mori S. A prospective randomized trial of extended cervical and superior mediastinal lymphadenectomy for carcinoma of the thoracic esophagus. Am J Surg. 1998 Jan;175(1):47-51. doi: 10.1016/s0002-9610(97)00227-4. PMID 9445239
- [Background] Watanabe H. [Necessity of cervical lymph node dissection by retrospective analysis of submucosal cancer in mid-thoracic esophagus]. Nihon Geka Gakkai Zasshi. 1997 Sep;98(9):733-6. Japanese. PMID 9370130
- [Background] Law SY, Fok M, Wong J. Pattern of recurrence after oesophageal resection for cancer: clinical implications. Br J Surg. 1996 Jan;83(1):107-11. doi: 10.1002/bjs.1800830134. PMID 8653330
- [Background] Medical Research Council Oesophageal Cancer Working Group. Surgical resection with or without preoperative chemotherapy in oesophageal cancer: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1727-33. doi: 10.1016/S0140-6736(02)08651-8. PMID 12049861
- [Background] Kelsen DP, Ginsberg R, Pajak TF, Sheahan DG, Gunderson L, Mortimer J, Estes N, Haller DG, Ajani J, Kocha W, Minsky BD, Roth JA. Chemotherapy followed by surgery compared with surgery alone for localized esophageal cancer. N Engl J Med. 1998 Dec 31;339(27):1979-84. doi: 10.1056/NEJM199812313392704. PMID 9869669
- [Background] Polee MB, Tilanus HW, Eskens FA, Hoekstra R, Van der Burg ME, Siersema PD, Stoter G, Van der Gaast A. Phase II study of neo-adjuvant chemotherapy with paclitaxel and cisplatin given every 2 weeks for patients with a resectable squamous cell carcinoma of the esophagus. Ann Oncol. 2003 Aug;14(8):1253-7. doi: 10.1093/annonc/mdg328. PMID 12881388
- [Background] Keresztes RS, Port JL, Pasmantier MW, Korst RJ, Altorki NK. Preoperative chemotherapy for esophageal cancer with paclitaxel and carboplatin: results of a phase II trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1603-8. doi: 10.1016/s0022-5223(03)00710-4. PMID 14666040
- [Background] Desoize B, Madoulet C. Particular aspects of platinum compounds used at present in cancer treatment. Crit Rev Oncol Hematol. 2002 Jun;42(3):317-25. doi: 10.1016/s1040-8428(01)00219-0. PMID 12050023
- [Background] Yamanaka H, Motohiro T, Michiura T, Asai A, Mori T, Hioki K. Nedaplatin and 5-FU combined with radiation in the treatment for esophageal cancer. Jpn J Thorac Cardiovasc Surg. 1998 Oct;46(10):943-8. doi: 10.1007/BF03217851. PMID 9847566
- [Background] Yoshioka T, Gamoh M, Shineha R, Ishibashi S, Shibata H, Suzuki T, Murakawa Y, Kato S, Shimodaira H, Kato S, Ishioka C, Kanamaru R. A new combination chemotherapy with cis-diammine-glycolatoplatinum (Nedaplatin) and 5-fluorouracil for advanced esophageal cancers. Intern Med. 1999 Nov;38(11):844-8. doi: 10.2169/internalmedicine.38.844. PMID 10563743
- See also: Related Info — http://www.sysucc.org.cn/